CLINICAL TRIAL: NCT03394170
Title: Pathogen Screening in OA Orthopaedic Surgical Patients
Status: Completed | Type: Observational
Sponsor: The Stone Research Foundation for Sports Medicine and Arthritis (Other)
Responsible Party: Sponsor
Other Study IDs: SRF-025
Record Dates: First submitted 2018-01-03; First posted 2018-01-09 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2018-01

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Osteoarthritis: Participants who are undergoing unicompartmental knee replacement will be considered OA status
  Interventions: Other: Collection of specimens prior to and during surgery
- Non-Osteoarthritis: Participants with an acute injury (occurring no more than 90 days prior to surgery) with no history of knee injury or surgery, will be considered "Non-OA" status
  Interventions: Other: Collection of specimens prior to and during surgery

INTERVENTIONS:
Other: Collection of specimens prior to and during surgery — Collection of specimens prior to and during surgery
  Other Names: Specimen collection

SUMMARY:
The purpose of this study is to screen orthopedic surgery patients with and without a diagnosis of osteoarthritis for the presence of 11 pathogens associated with periodontal disease (PD) from a collection of oral rinse, synovial fluid and their synovium. The investigators hypothesize that there is a correlation between the presence of specific oral pathogens in saliva, synovial fluid and synovial tissue with clinical diagnosis of OA.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is the most common form of arthritis, affecting over 27 million people in the US. Rheumatoid arthritis (RA), a less common form of arthritis, is believed to differ from OA in its etiology, however both result in breakdown of cartilage. Studies have reported the association between chronic or adult periodontal disease (PD), Porphyromonas gingivalis (P. gingivalis), a gram-negative anaerobic bacterium, and rheumatoid arthritis (RA). Whether or not there is an infectious component of osteoarthritis is of significant interest.

The purpose of this study is to screen orthopedic surgery patients with and without a diagnosis of osteoarthritis for the presence of 11 pathogens associated with PD from a collection of oral rinse, synovial fluid and their synovium. The investigators hypothesize that there is a correlation between the presence of specific oral pathogens in saliva, synovial fluid and synovial tissue with clinical diagnosis of OA.

If an association between OA disease status and the presence of one or more pathogens can be confirmed, further studies can be undertaken to investigate the causative nature of oral pathogens in the clinical manifestation of OA, and eventually may lead to development of targeted therapies to prevent or slow the progression of OA.

This study will recruit 50 patients with indications for knee surgery, who fit the inclusion/exclusion criteria. Prior to surgery, patients will undergo an Institutional Review Board (IRB) approved informed consent process for in vitro cellular and biochemical characterization of their tissue. Two discreet populations, essentially normal knees and confirmed osteoarthritic knees will be studied. All patients will provide specimens for analysis, to identify the presence of oral pathogens in each participants saliva, synovial fluid and synovium.

Evaluation will include identifying the type and concentration of the following perio-pathogenic bacteria that are known to cause periodontal disease:

* Aggregatibacter actinomycetemcomitans
* Campylobacter rectus
* Capnocytophaga species (gingivalis, ochracea, sputigena)
* Eikenella corrodens
* Eubacterium nodatum
* Fusobacterium nucleatum/periodonticum
* Parvimonas micra
* Porphyromonas gingivalis
* Prevotella intermedia
* Tannerella forsythia
* Treponema denticola

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature (as evidenced by x-ray)
* Aged 18 years or over
* Patient will be undergoing orthopaedic surgery
* If patient is "Non-OA," patient has no history of previous injury / surgery to operative joint
* Patient is able to understand the requirements of the study, abide by the restrictions, and return for all required examinations and treatments.
* Patient is able to give written informed consent

Exclusion Criteria:

* A clinical diagnosis of inflammatory arthritis made by history, examination or serology.
* An active or latent infection of the affected knee joint or any other systemic infection currently under treatment or treated within the previous 3 months.
* A history of chronic alcohol or drug abuse during the six months prior to the study.
* Clinically documented acute or unstable concomitant disease, other than the condition to be treated in this study that might affect make it difficult to interpret the patient's cartilage composition (i.e. renal, hepatic, cardiac, endocrine, hematologic, autoimmune, metabolic bone, crystal deposition, severe degenerative joint, neoplastic diseases).
* Systemic administration, within twenty days prior to the procedure, of any type of corticosteroids, antineoplastic, immunostimulating or immunosuppressant agents.
* Patients with a medical condition that interferes with their ability to participate in surgery or rehabilitation program.
* Participation in any other investigational drug or device trial during the 30 days prior to screening visit or who will receive such a drug or device during the course of this study.
* Pregnant females.
* Subject's unable or unwilling to comply with the protocol or scheduled appointments.
* Subject's unable to provide informed consent.
* Subject's unable to understand verbal and/or written English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending The Stone Clinic for knee surgery as a result of a recent sports injury or known osteoarthritis can be considered if they fit the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Evidence of oral pathogens in knee joint | 2 weeks
  Evidence of specified oral pathogens in the synovial fluid and/or tissue

CONTACTS AND LOCATIONS:
Overall Officials: Kevin R Stone, MD, Principal Investigator — Foundation for Sports Medicine & Arthritis Research (Stone Research Foundation)
Locations (1):
- Stone Research Foundation, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No